CLINICAL TRIAL: NCT04704726
Title: Examining Essentialistic Beliefs About Food
Status: Completed | Type: Observational
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Ciaran Forde, Senior Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Other Study IDs: 2020-05-045
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project seeks to test whether people maintain essentialistic beliefs about food (foods as having immutable underlying 'essences' that contribute to the food's attributes and properties). Currently, there are studies on essentialistic beliefs on topics such as: race, genes, and natural objects. However, there is limited research applying the concept of essentialism to food. In addition, in food studies, participants' perception and acceptability of foods were being explored but what remains unknown is whether they have any degree of essentialistic beliefs towards food which influences their perception and acceptability of food.

Therefore, the aim of this study is to gain in-depth knowledge and understanding on whether people maintain essentialistic beliefs about food, and determine whether these beliefs may be associated with attitudes and expectations of foods that vary in their levels of processing.

DETAILED DESCRIPTION:
Objectives:

1. To gain in-depth knowledge and understanding on whether people maintain essentialistic beliefs about food (foods as having immutable underlying 'essences' that contribute to the food's attributes and properties).
2. To determine whether these beliefs may be associated with attitudes and expectations of foods that vary in their levels of processing.
3. To explore the perceptions of essentialistic transference: The belief that the essence of a food is transferred to a person who consumes the food, which manifests the properties of the food in the consumer (E.g., the belief that people who have a diet of eating fast-running animals are also fast runners).

Study Design:

This study involves 2 parts: Study 1A & Study 1B.

Study 1A:

300 participants in Singapore, aged between 21-65 years old will be recruited to do an online survey on Qualtrics. Participants would first rate their baseline appetite before proceeding to the survey. For this study, the food categories will be: Milk, Rice, Carrot and Chicken. There will be a total of 7 different kinds of foods varying in the levels of processing per category and the images of these foods will be presented in a randomized order. Participants will rate their perceptions of the properties of foods (e.g. nutritiousness, naturalness, familiarity, liking, taste, stereotypical trait, and processing) on a scale that ranges from "Not at all" to "Very much".

After rating their perceptions of the properties of foods, participants will complete questionnaires measuring: Essentialistic beliefs about food (EFS: 6-point scale from "Strongly Disagree" to "Strongly Agree"), perceptions of essentialistic transference (ETS: 6-point scale with 2 opposite traits as anchors e.g. "Very Irritable" to "Very good-natured"), nutrition knowledge (NKS: 6-point scale from "Strongly Disagree" to "Strongly Agree"), importance of food naturalness (FNS: 6-point scale from "Strongly Disagree" to "Strongly Agree") and consumers' fears towards food technology (FTNS: 7-point scale from "Strongly Disagree" to "Strongly Agree").

Study 1B:

300 participants in Singapore, aged between 21-65 years old will be recruited to do an online survey on Qualtrics. Participants would first rate their baseline appetite before proceeding to the survey. For this study, the food categories will be: Fish, Orange, Napa Cabbage, Peanut and Beef. There will be a total of 7 different kinds of foods varying in the levels of processing per category and 2 foods-in-name (e.g. Vuna and Impossible burger), and the images of these foods will be presented in a randomize order. Participants will rate their perceptions of the properties of foods (e.g. nutritiousness, naturalness, familiarity, liking, taste, stereotypical trait, and processing) on a scale that ranges from "Not at all" to "Very much".

After rating their perceptions of the properties of foods, participants will complete questionnaires measuring: Essentialistic beliefs about food (EFS: 6-point scale from "Strongly Disagree" to "Strongly Agree"), perceptions of essentialistic transference (ETS: 6-point scale with 2 opposite traits as anchors e.g. "Very Irritable" to "Very good-natured"), nutrition knowledge (NKS: 6-point scale from "Strongly Disagree" to "Strongly Agree"), importance of food naturalness (FNS: 6-point scale from "Strongly Disagree" to "Strongly Agree") and consumers' fears towards food technology (FTNS: 7-point scale from "Strongly Disagree" to "Strongly Agree").

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old

Exclusion Criteria:

* None

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the general public of Singapore aged between 21-65 years old, through Dynata (a market research company).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Consumers' perceptions of food | Baseline measure
  Participants will be shown images of different kinds of foods varying in the levels of processing and they will rate their perceptions of the properties of foods (e.g., nutritiousness, naturalness, familiarity, liking, taste, stereotypical trait, and processing) on a scale that ranges from "Not at all" to "Very much".
Essentialistic beliefs about food (food as having immutable underlying 'essences' that contribute to the food's attributes and properties) | Baseline measure
  The essentialistic beliefs about food will be measured by a scale that we developed: Essentialism of Food Scale (EFS): 6-point scale from "Strongly Disagree" to "Strongly Agree".
Perceptions of essentialistic transference | Baseline measure
  Perceptions of essentialistic transference refers to the belief that the essence of a food is transferred to a person who consumes the food, which manifests the properties of the food in the consumer (e.g., the belief that people who have a diet of eating fast-running animals are also fast runners). It will be measured by a scale that we developed: Essentialistic Transference Scale (ETS): 6-point scale with 2 opposite traits as anchors e.g. "Very Irritable" to "Very good-natured"
Nutrition knowledge | Baseline measure
  Nutrition knowledge will be measured by the Nutrition Knowledge scale (NKS): 6-point scale from "Strongly Disagree" to "Strongly Agree".
Perception towards the importance of food naturalness | Baseline measure
  Importance of food naturalness will be measured by the Food Naturalness Scale (FNS): 6-point scale from "Strongly Disagree" to "Strongly Agree".
Consumers' fears towards food technology | Baseline measure
  Consumers' fears towards food technology will be measured by the Food Technology Neophobia Scale (FTNS): 7-point scale from "Strongly Disagree" to "Strongly Agree".

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Cheon, PhD, Principal Investigator — Bobby_Cheon@sics.a-star.edu.sg
Locations (1):
- Singapore, Singapore, Singapore